CLINICAL TRIAL: NCT03503929
Title: A Pilot Study Evaluating the Feasibility and Usability of the LaparoGuard System During Laparoscopic Surgical Procedures
Brief Title: Feasibility and Usability of LaparoGuard
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mariner Endosurgery (Industry)
Collaborators: Hamilton Health Sciences Corporation (Other); Federal Economic Development Agency for Southern Ontario (FedDev Ontario) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: LAP-PRO-001
Record Dates: First submitted 2018-01-25; First posted 2018-04-20 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Laparoscopic Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Open label, prospective, single site, multi-investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LaparoGuard System (Other): All patients receiving laparoscopic surgery, candidates for prolonged time under anesthesia, and are admitted for gynecological, urological or general surgery procedures who consent to use of the LaparoGuard System.
  Interventions: Device: LaparoGuard System

INTERVENTIONS:
Device: LaparoGuard System — Adjunctive safety system for laparoscopic surgery

SUMMARY:
LaparoGuard is intended as an adjunctive safety system for laparoscopic surgery. The system allows surgeons to virtually annotate a safe anatomical volume inside the body cavity of the patient during a laparoscopic surgery. The surgeon then receives notification throughout the procedure whenever a tracked rigid instrument has exited that volume. This open label, prospective, feasibility, single site, multi-investigator trial will evaluate the feasibility and usability of the LaparoGuard system during laparoscopic surgical procedures.

DETAILED DESCRIPTION:
PHASE 1) LaparoGuard will be used as an adjunctive tool for maintaining safety during procedures performed by expert surgeons. The pre-operative instructions for use will be evaluated along with ease of procedural setup, as reported by pre-operative nurses. The intraoperative instructions for use will be evaluated along with system usability, as reported by the expert surgeons. The perceived clinical utility will be judged by expert surgeons. Postoperatively, the system data will be reviewed. This phase will include 4-6 subjects.

PHASE 2) Novice surgeons will conduct procedures alongside expert surgeons. Expert surgeons will establish the safe zone. LaparoGuard will record all deviations, speed and smoothness of tip movements. The training utility of LaparoGuard will be assessed by both the expert and novice surgeons. This phase will include 4-6 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing routine laparoscopic procedures. Examples include (non-exhaustive): operative laparoscopy, appendectomy, cholecystectomy, colon resection, inguinal or diaphragmatic hernia repairs.
* Ability to read and understand English
* Consent to use of the LaparoGuard system in their procedure (18 yrs or older)

Exclusion Criteria:

* Unwilling to sign informed consent
* Simple diagnostic laparoscopy (can be included if conversion to operative laparoscopy)
* Surgeries which require conversion to laparotomy for patient safety reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-21 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Procedural Success | Intraoperative
  For each surgical procedure conducted, the case will be defined as a technical success if: the surgical team is able to complete the procedure without needing to turn off the LaparoGuard system. Failure will be if the operator deems it necessary to stop utilizing the LaparoGuard system and resort to the standard (non-annotated) endoscopic camera feed. Potential reasons for doing so may be device reporting errors, such as the LaparoGuard system consistently incorrectly reporting that a surgical tool has exited the safe zone.
  In emergency situations, such as changes in medical condition unrelated to use of the LaparoGuard system, the operator may also deem it necessary to resort to the standard-of-care; however, these situations will not be judged as failures and the case data will be utilized for study purposes up until that point.

SECONDARY OUTCOMES:
Pre-operative LaparoGuard system setup time | Baseline
  The amount of time taken to setup the LaparoGuard system by the surgical nurses will be recorded
Usability reported pre-operatively by nurses | Baseline
  Following setup of the LaparoGuard system preoperatively, but prior to bringing the patient into the surgical suite, study staff will conduct a short interview with the surgical nurses to evaluate their comfort and ease with the system setup procedures. If any use errors or confusion were observed by the study staff, these shall be discussed in depth. Comments reported by the nurses on difficulties encountered and potential simplifications to the procedures will be recorded.
Safe zone deviations | Intraoperative
  The total number of safe zone deviations as well the total time each instrument was outside the safe zone will be tracked and evaluated.
Usability reported post-operatively by surgical team | Intraoperative
  Following completion of each surgical procedure, study staff will conduct a short interview with the surgical team to evaluate the ability of the team to interpret the LaparoGuard output, the safe zone and respond to any information provided by system.
Clinical utility reported by expert surgeons | 2 months
  Following the completion of all 10 cases, study staff will conduct interviews with the expert surgeons to evaluate their perceived clinical utility of the LaparoGuard system. A qualitative discussion will held around the particular clinical situations in which LaparoGuard may be most useful. Study staff will also record any potential insights by the surgeons on future features which may be incorporated to improve the clinical utility of LaparoGuard.
Training utility reported by novice and expert surgeons | 2 months
  Following the completion of all 10 cases, study staff will conduct interviews with the expert and novice surgeons to evaluate their perceived training utility of the LaparoGuard system. Quantitative rating scales will be used and qualitative discussion will held around the particular training situations in which LaparoGuard may be most useful. Study staff will also record any potential insights by the expert or novice surgeons on future features which may be incorporated to improve the training utility of LaparoGuard.

CONTACTS AND LOCATIONS:
Overall Officials: Niv Sne, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No